CLINICAL TRIAL: NCT03563872
Title: Enhancing Systems of Care to Improve Hypertension Guideline Implementation to Communities With Health Disparities
Brief Title: Enhancing Systems of Care to Improve Hypertension Guideline Implementation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Joseph Miller, MD, Senior Staff, Henry Ford Health System
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 13455
Record Dates: First submitted 2018-06-10; First posted 2018-06-20 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Hypertension
Keywords: hypertension; team-based; guidelines; implementation
MeSH Terms: conditions — Hypertension | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Team-based care
  Interventions: Other: Active Comparator
- Intervention (Experimental): Enhanced team-based care
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Enhancements to team-based care include clinical decision support and improved protocols for telehealth prescribing.
  Arms: Intervention
Other: Active Comparator — Usual, team-based care
  Arms: Active Comparator

SUMMARY:
This study is a prospective cluster randomized trial testing a systems-level strategy to implement current American Heart Association hypertension guidelines in African American communities at risk for cardiovascular related health disparities. The trial will take place within an integrated health system serving Detroit and will assess blood pressure control over one year's time.

DETAILED DESCRIPTION:
The trial will randomize 12 clinics within the Henry Ford Health System to two arms. The first arm will be comparison clinics that continue to use existing team-based strategies for hypertension management. The second arm will be intervention clinics. These clinics will have enhancements to existing team-based hypertension management. The first enhancement is clinical decision support based in the electronic health record. The second enhancement is improved protocols to implement telehealth prescribing that is nurse-led.

The trial will enroll participants through an urban emergency department. Participants will be assigned to one of these 12 clinics and continue study activities for 1 year. Clinicians at the clinics will manage blood pressure. Study specific visits will occur at 3, 6, 9, and 12 months. Primary outcome assessment is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) African Americans
* Lacks established primary care for BP management
* History of HTN
* SBP ≥ 140 mmHg

Exclusion Criteria:

* Pregnancy
* Need for hospitalization from ED
* Serious comorbid conditions
* Alcohol or drug dependence
* Suspected resistant HTN
* Anticipated poor-adherence to study designated primary care clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure | 12 months
  mean change

SECONDARY OUTCOMES:
Therapeutic Intensity | 12 months
  Calculated therapeutic intensity score
Change in systolic blood pressure | 6 months
  mean change
Change in diastolic blood pressure | 12 months
  mean change
Treatment Congruence | 12 months
  Proportion of clinical encounters in which treatment is congruent with guidelines

OTHER OUTCOMES:
Cost effectiveness | 12 months
  within trial cost and long-term projected costs compared to QALY

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided